CLINICAL TRIAL: NCT07062770
Title: Assessment of Circuit Rebreathing During Continuous Positive Airway Pressure (CPAP) Therapy
Brief Title: Assessment of Circuit Rebreathing During CPAP Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: Sleep Res, Inc. (Unknown)
Responsible Party: Principal Investigator, Atqiya Aishah, Ph.D., Postdoctoral Research Fellow, Brigham and Women's Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Other
Other Study IDs: 2025P000798
Record Dates: First submitted 2025-05-27; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Obstructive Sleep Apnea (OSA)
Keywords: Obstructive sleep apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Intervention Model Description: Subjects will perform 1 in-lab sleep study visit consisting of an evening wake session followed by an overnight sleep study.
  Subjects will receive randomized sequences of 11 conditions (varying in exhaust flow and PAP levels) during the evening and sleep portions of the night.
Who Masked: Participant
Masking Description: The exhaust flow and PAP level conditions will be blinded for the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (11):
- 5 cmH2O with 35L/s (Experimental): 35 L/s exhaust flow with 5 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 5 cmH2O with 23L/s (Experimental): 23 L/s exhaust flow with 5 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 5 cmH2O with 18L/s (Experimental): 18 L/s exhaust flow with 5 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 5 cmH2O with 13L/s (Experimental): 13 L/s exhaust flow with 5 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 5 cmH2O with 8L/s (Experimental): 8 L/s exhaust flow with 5 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 0 cmH2O with 35L/s (Placebo Comparator): 35 L/s exhaust flow with 0 cmH₂O PAP
  Interventions: Other: Mask exhaust port flow
- 10 cmH2O with 35L/s (Experimental): 35 L/s exhaust flow with 10 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 10 cmH2O with 23L/s (Experimental): 23 L/s exhaust flow with 10 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 10 cmH2O with 18L/s (Experimental): 18 L/s exhaust flow with 10 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 10 cmH2O with 13L/s (Experimental): 13 L/s exhaust flow with 10 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow
- 10 cmH2O with 8L/s (Experimental): 8 L/s exhaust flow with 10 cmH₂O PAP
  Interventions: Device: Continuous positive airway pressure (CPAP); Other: Mask exhaust port flow

INTERVENTIONS:
Device: Continuous positive airway pressure (CPAP) — Subjects will be administered either 0, 5 or 10 cmH2O
  Arms: 10 cmH2O with 13L/s; 10 cmH2O with 18L/s; 10 cmH2O with 23L/s; 10 cmH2O with 35L/s; 10 cmH2O with 8L/s; 5 cmH2O with 13L/s; 5 cmH2O with 18L/s; 5 cmH2O with 23L/s; 5 cmH2O with 35L/s; 5 cmH2O with 8L/s
Other: Mask exhaust port flow — Subjects will be administered varying levels of exhaust flow: 35, 23, 18, 13 and 8 L/s

SUMMARY:
The goal of this research is to better understand how different CPAP mask designs affect airflow and rebreathing of exhaled carbon dioxide (CO₂) during sleep in individuals with obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
To understand the existence and severity of circuit rebreathing during treatment with continuous positive airway pressure (CPAP) using different sizes of the exhaust ports in individuals with obstructive sleep apnea (OSA).

Flow-adjusted end-tidal oxygen (PetO2) and carbon dioxide (PetCO2) will be assessed to determine the magnitude of hypoxic load during both wakefulness and sleep. To systematically assess these conditions, the conditions were defined as follows:

* 5A: 35 L/s exhaust flow with 5 cmH₂O PAP
* 5B: 23 L/s exhaust flow with 5 cmH₂O PAP
* 5C: 18 L/s exhaust flow with 5 cmH₂O PAP
* 5D: 13 L/s exhaust flow with 5 cmH₂O PAP
* 5E: 8 L/s exhaust flow with 5 cmH₂O PAP
* 0P: 35 L/s exhaust flow with 0 cmH₂O PAP
* 10A: 35 L/s exhaust flow with 10 cmH₂O PAP
* 10B: 23 L/s exhaust flow with 10 cmH₂O PAP
* 10C: 18 L/s exhaust flow with 10 cmH₂O PAP
* 10D: 13 L/s exhaust flow with 10 cmH₂O PAP
* 10E: 8 L/s exhaust flow with 10 cmH₂O PAP Primary endpoint is to evaluate the effect of exhaust flow on flow-adjusted average inspired oxygen fraction (FiO₂) during (1) wakefulness and (2) sleep between 5B vs. 5D.

ELIGIBILITY:
Inclusion Criteria:

* Moderate to severe OSA (AHI>20)
* Self-reported CPAP users or have previously used CPAP
* Self-reported holding pressure of maximum 13 cmH2O (if known)
* Age: 21-70
* BMI: 18-40 kg/m2

Exclusion Criteria:

* Self-reported severe mouth-breathing
* Requirement for nocturnal supplemental oxygen or other ventilatory support
* Severe cardiovascular or pulmonary disease
* Any unstable or acute medical condition
* Any additional sleep disorder, including insomnia, except for OSA.

Ages: 21 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2025-05-27 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Change in flow-adjusted average inspired oxygen fraction (FiO₂) during wake. | through study completion, an average of 1 year
  Difference in FiO2 between 23L/s vs 13L/s exhaust flow at 5 cmH2O PAP.
Change in flow-adjusted average inspired oxygen fraction (FiO₂) during sleep. | through study completion, an average of 1 year
  Difference in FiO2 between 23L/s vs 13L/s exhaust flow at 5 cmH2O PAP.

SECONDARY OUTCOMES:
Impact on hypoxic burden during sleep. | through study completion, an average of 1 year
  Difference in hyboxic burden between 23L/s vs 13L/s exhaust flow at 5 cmH2O PAP.

CONTACTS AND LOCATIONS:
Overall Officials: Atqiya Aishah, PhD, Principal Investigator — Harvard Medical School & Brigham and Women's Hospital
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified subject data will be available upon request.